CLINICAL TRIAL: NCT02594189
Title: Influenza A H3N2 Human Challenge Study in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 160008; 16-I-0008
Record Dates: First submitted 2015-10-31; First posted 2015-11-03 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2017-11-01

CONDITIONS: Determine Minimally to Moderately Infective Dose (MMID) of Influenza A H3N2
Keywords: Influenza A; H3N2; Challenge Model; Influenza; Human Challenge
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- 1 (Other): The human challenge virus will be administered intranasally to each participant using a nasal sprayer. A total volume of up to 2mL of virus will be administered.
  Interventions: Other: Live recombinantly derived A/Bethesda/MM1/H3N2 virus

INTERVENTIONS:
Other: Live recombinantly derived A/Bethesda/MM1/H3N2 virus — The human challenge virus will be administered intranasally to each participant using a nasal sprayer. A total volume of up to 2mL of virus will be administered.

SUMMARY:
Background:

Influenza A H3N2 is a flu virus. Symptoms include fever, cough, and runny nose. It can also be more serious. Researchers want to know more about how influenza causes disease in people. They hope to develop new vaccines and treatments for flu infection.

Objective:

To find the smallest amount of Influenza A H3N2 virus that causes a mild to moderate flu infection in healthy people. Also, to study the body s immune response to this virus and how the infection develops.

Eligibility:

Healthy people ages 18 50 who are:

Non-smokers or non-habitual smokers

Willing to not smoke for at least 9 days

Design:

Participants will be screened under NIAID protocol #11-I-0183

Participants will stay at an isolation unit at the clinic for at least 9 days. They will remain in the isolation unit except for study-specific activities.

The influenza virus will be sprayed into the nose.

Participants will be monitored 24 hours a day. They will have tests, including:

Medical history

Physical exam

Daily questionnaires about symptoms

Blood and urine tests

Nasal wash and swab: A small tube of salt water is placed in the nose to wash it. It then collects the

fluid. Or the inside of the nose is rubbed with a swab.

ECG: Measures the heart s electrical signals

ECHO: Sound waves take pictures of the heart

PFTs/Spirometry: They will blow into a machine that measures the air they blow.

Participants will be discharged after they test negative for influenza A.

Participants will return to the clinic for 4 follow-up visits over 8 weeks. They may complete questionnaires at home.

DETAILED DESCRIPTION:
The high morbidity and mortality associated with both pandemic and seasonal influenza, and the anticipation of future influenza pandemics, puts influenza front and center in infectious disease research. Because the natural history and pathogenesis of human influenza has not been well characterized and cannot be adequately studied in animal models or with current in vitro techniques, important questions about influenza pathogenesis can only be approached through human challenge studies.

Although studies of influenza in healthy volunteers have played an important role in addressing aspects of the natural history of influenza disease and developing novel antivirals, prior to recently these important studies had not been performed in the US in over a decade. The H1N1 challenge studies we have performed since 2012 have sought to improve upon the studies done in the past and address many of the limitations due to the scope of the studies and/or the scientific techniques available at that time. We have successfully developed an H1N1 model that had been used to address important questions regarding correlates of protection and is now being implemented to develop new drugs and vaccines. We hope to develop H3N2 models that can be just as useful.

The primary objective of this study is to determine the dose of influenza A H3N2 human challenge virus that will induce a mild to moderate uncomplicated influenza infection in healthy volunteers. This protocol will examine some of the basic questions that remain unanswered regarding the pathogenesis of H3N2 influenza in humans, namely, a detailed clinical and immunological characterization of uncomplicated influenza viral pathogenesis in healthy adult volunteers.

Secondary objectives will evaluate clinical disease, length of viral shedding, and pathogenesis in those with influenza infection including identification of clinical markers of the disease. Notably, the exploratory objectives will seek to discover viral factors necessary for human infection/adaptation and to evaluate host immune response, viral replication, viral fitness, and the intrahost evolution.

Collaboration between NIAID investigators and outside scientists will generate opportunities to further develop and expand areas of clinical influenza research based on the proposed H3N2 challenge model.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Greater than or equal to 18 and less than or equal to 50 years of age.
2. Agrees to not use tobacco products during participation in this study.
3. Willingness to remain in isolation for the duration of viral shedding (at a minimum 9 days) and to comply with all study requirements.
4. A female participant is eligible for this study if she is not pregnant or breastfeeding and meets 1 of the following criteria:

   * Of nonchildbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in more than or equal to 1 year).
   * Of childbearing potential but agrees to practice effective contraception or abstinence for 4 weeks prior to and 8 weeks after administration of the influenza challenge virus. Acceptable methods of contraception include 1 or more of the following: 1) male partner who is sterile prior to the female participant s entry into the study and is the sole sexual partner for the female participant; 2) implants of levonorgestrel; 3) injectable progestogen; 4) an intrauterine device with a documented failure rate of <1%; 5) oral contraceptives; and 6) double barrier methods including diaphragm or condom with a spermicide.
5. Willing to have samples stored for future research.
6. Pre-challenge serum hemaglutination-inhibition titer against the challenge strain of less than 1:40.
7. HIV uninfected.

EXCLUSION CRITERIA:

1. Presence of self-reported or medically documented significant medical condition including but not limited to:

   1. Chronic pulmonary disease (e.g., asthma, emphysema).
   2. Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
   3. Chronic medical conditions requiring close medical follow-up or hospitalization during the past 5 years (e.g., insulin-dependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
   4. Immunosuppression or ongoing malignancy.
   5. Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
   6. Post infectious or post vaccine neurological sequelae.
2. Have close or household (i.e., share the same apartment or house) high-risk contacts including but not limited to:

   1. Persons more than or equal to 65 years of age.
   2. Children less than or equal to 5 years of age.
   3. Residents of nursing homes.
   4. Persons of any age with significant chronic medical conditions such as:

      * Chronic pulmonary disease (e.g., asthma).
      * Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
      * Contacts who required medical follow-up or hospitalization during the past 5 years because of chronic medical conditions (e.g., insulindependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
      * Immunosuppression or cancer.
      * Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
      * Persons who are receiving long-term aspirin therapy.
      * Women who are pregnant, trying to become pregnant, or breastfeeding.
3. Individual with body mass index (BMI) less than or equal to 18.5 and more than 40.
4. Smokes more than 4 cigarettes or other tobacco products on weekly basis.
5. Complete blood count (CBC) with differential outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
6. Chemistries in the acute care, mineral, and/or hepatic panels, and/or any of the following: lactate dehydrogenase, uric acid, creatine kinase, and total protein outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
7. Urinalysis outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
8. Clinically significant abnormality as deemed by the PI on electrocardiogram (EKG)
9. Clinically significant abnormality as deemed by the PI on echocardiographic testing (ECHO).
10. Clinically significant abnormality as deemed by the PI on the Pulmonary Function Test (PFT).
11. Recent acute illness within 1 week of admission to the isolation facility.
12. Known allergy to treatments for influenza (including but not limited to oseltamivir, nonsteroidals).
13. Known allergy to 2 or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
14. Receipt of blood or blood products (including immunoglobulins) within 3 months prior to enrollment.
15. Receipt of any unlicensed drug within 3 months or 5.5 half-lives (whichever is greater) prior to enrollment.
16. Receipt of any unlicensed vaccine within 6 months prior to enrollment.
17. Self-reported or known history of current alcoholism or drug abuse, or positive urine/serum test for drugs of abuse (i.e., amphetamines, cocaine, benzodiazepines, opiates, or metabolites, but not THC or metabolites).
18. Self-reported or known history of psychiatric or psychological issues deemed by the PI to be a contraindication to protocol participation
19. Known close contact with anyone known to have influenza in the past 7 days.
20. Any condition that, in the judgment of the PI, is a contraindication to protocol participation or impairs the volunteer s ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2015-10-31; Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Determine the minimally to moderately infective dose (MMID) of influenza A H3N2 human challenge virus, defined as the dose that induces uncomplicated mild to moderate influenza infection in at least 60% of healthy volunteers. | 2 yr

SECONDARY OUTCOMES:
Evaluate clinical disease, identify clinical markers, and observe initiation of shedding, length of shedding, and pathogenesis in participants with influenza infection. | 1yr

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Carrat F, Vergu E, Ferguson NM, Lemaitre M, Cauchemez S, Leach S, Valleron AJ. Time lines of infection and disease in human influenza: a review of volunteer challenge studies. Am J Epidemiol. 2008 Apr 1;167(7):775-85. doi: 10.1093/aje/kwm375. Epub 2008 Jan 29. PMID 18230677
- [Background] Anderson MJ, Heath RB. Cell mediated immunity in experimental influenza and parainfluenza infection. Dev Biol Stand. 1977 Jun 1-3;39:379-83. PMID 203505
- [Background] Brown TA, Murphy BR, Radl J, Haaijman JJ, Mestecky J. Subclass distribution and molecular form of immunoglobulin A hemagglutinin antibodies in sera and nasal secretions after experimental secondary infection with influenza A virus in humans. J Clin Microbiol. 1985 Aug;22(2):259-64. doi: 10.1128/jcm.22.2.259-264.1985. PMID 4031039
- [Derived] Han A, Czajkowski LM, Donaldson A, Baus HA, Reed SM, Athota RS, Bristol T, Rosas LA, Cervantes-Medina A, Taubenberger JK, Memoli MJ. A Dose-finding Study of a Wild-type Influenza A(H3N2) Virus in a Healthy Volunteer Human Challenge Model. Clin Infect Dis. 2019 Nov 27;69(12):2082-2090. doi: 10.1093/cid/ciz141. PMID 30770534